CLINICAL TRIAL: NCT04608084
Title: Platelet Rich Plasma Eye Drops for Treatment of Ocular Surface Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Allan Slomovic, M.D, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-5033.0
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Ocular Surface Disease; Dry Eye Syndromes
Keywords: Dry eye syndrome; Platelet rich plasma; ocular surface disease; Autologous serum
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Participant with moderate to sever ocular surface disease will be treated with autologous platelet rich plasma eye drops
  Interventions: Biological: Autologous platelet rich plasma eye drops

INTERVENTIONS:
Biological: Autologous platelet rich plasma eye drops — Participant own blood is used for the preparation of Autologous platelet rich plasma eye drops

SUMMARY:
The purpose of this study is to evaluate prospectively the efficacy of topical administration of autologous platelet rich plasma as monotherapy for the treatment of symptoms and clinical signs in cases affected by moderate to severe forms of ocular surface disease

DETAILED DESCRIPTION:
Background Ocular Surface Disease (OSD) is a multifactorial disease of the ocular surface and tears that produce symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface. It is accompanied by increased osmolarity of the tear film and inflammation of the ocular surface. The prevalence of Ocular surface disease reported in the literature up to 30% of the elderly population. There are two main mechanisms that explain this ocular surface dysfunction: aqueous deficiency and excessive evaporation of the tear film. The aqueous deficient dry eye disease is characterized by an insufficient volume of tears due to dysfunction of the lacrimal glands and obstruction of the lacrimal ducts. This mechanism is also related to autoimmune diseases such as Sjogren's syndrome, Lupus, and Rheumatoid arthritis. Meibomian gland dysfunction, eyelid problems (infrequent blinking, entropion, ectropion) are typical causes of evaporative dry eye. Poor tear film quality is the result of tear hyperosmolarity and goblet cell mucin deficiency. Ocular surface disease can also arise as iatrogenic complication after external or internal ocular surgery, laser treatment, radiation, chemotherapy or ocular medications.

Treating ocular surface diseases can be challenging and treatment usually depends on the underlining etiology and can be divided into medical treatment and surgical solutions. Non preserved artificial tears are usually the first line treatment for OSD associated with aqueous deficiency and anti-inflammatory drops like steroids, lifitegrast 5% (Xiidra-shire) and cyclosporin 0.05% (Restasis - allergan) often accompanied for treating the underling inflammatory process, However, none of these treatment includes essential tear components such as growth factors, vitamins, and immunoglobulins.

Hemoderivatives drops such as autologous serum (AS) have been recommended for the treatment of several ocular surface disturbances, such as Sjögren's syndrome-related tear deficiency, non-Sjögren's tear deficiency associated with graft-versus-host disease, neurotrophic keratitis, persistent epithelial defects, superior limbic keratoconjunctivitis, as well as a supportive measure in ocular surface reconstruction.

Platelet rich plasma (PRP) has been reported as successful treatments for moderate to severe OSD caused by dry eye, presenting advantages over AS due to its richer concentration of growth factors, anti-inflammatory cytokines, and other platelet derivatives. The high concentration of platelets obtained through a relatively simple process, which requires minimal manipulation and no addition of any other substance.

studies have shown that these components help in the proliferation, migration, and differentiation of corneal epithelial cells, which is beneficial for the required ocular surface restoration in moderate to severe forms of OSD

Investigated product Name Autologous Platelet rich plasma Indications Ocular surface diseases

Preparation and handling

For preparation of autologous PRP eye drops, dedicated closed system "ECLIPSE PRP PLATELET PREPARATION SYSTEM" which is health Canada approved, will be used.

peripheral blood from participants own antecubital vein will be collected into 12 mL tube, then it will be centrifuged at 580× g for 8 min at room temperature in an Eclipse System centrifuge "ECLIPSE EASY SPIN".

The whole column of PRP will be collected after centrifugation, avoiding the buffy coat that contains the leukocytes, using a sterile 10ml syringe, then the product is divided into 10 vials of 1ml each through a closed system. The vials will be given to the patient in a sealed box with ice packs.

Methodology Patient selection Inclusion criteria: Potential patients diagnosed with OSD will be identified at Dr. Slomovic's Cornea clinic at Toronto Western Hospital. Patients will be included when the fluorescein corne-conjunctival staining score is 5 or more as determined by NEI/Industry Grading System17 and OSDI questionnaire score of 20 or more, after treatment with non-preserved artificial tears 4/day for at least 1 month.

Patients will be excluded when they are under the age of 18 years or incapacitated patients.

If both eyes in one patient meet the inclusion criteria, the eye with higher corneal fluorescein staining score will be enrolled and analyzed for the study (although both eyes will be subject to treatment). If both eyes have the same score, the right eye will be enrolled.

For the purpose of this study, 100 participants will be enrolled. Main steps of the study Step 1: Recruitment, consenting the participant Step 2: Baseline evaluation and PRP preparation visit Step 3: Treatment effect monitoring visit, 6 weeks post treatment initiation Step 4: Follow-up visit, 6 weeks post treatment completion

Recruitment, consenting the participant Following clinical evaluation, the ophthalmologist decides if the patient meets the study criteria. If the prospective participant is eligible and interested in the project, a qualified member of the team will explain the benefits and risks of the trial and obtain informed consent, the patient will have the right to refuse participating in the study and will have time to ask questions regarding the study. Patient could advice his family and friends before signing the informed consent. patient will have no time limit for signing the informed consent.

Baseline, 6-week and 12 weeks assessment Prior to baseline assessment, informed consent will be obtained.

At baseline, after 6 weeks of treatment and 6 weeks post finishing the treatment. The following will be examined:

1. Subjective dry eye symptoms as assessed by the Ocular Surface Disease Index (OSDI) questionnaire
2. The noninvasive tear film break-up time (TFBUT)
3. Aqueous tear secretion as evaluated by Schirmer I test
4. Corneo-conjunctival staining scores graded by NEI/Industry Grading System after 1% fluorescein dye staining
5. Keratograph 5M (Oculus, Wetzlar, Germany)
6. Tear film osmolarity with a lab-on-a-chip technique (TearLab; TearLab Corporation, San Diego, CA, USA)
7. Central corneal sensitivity test by Cochet-Bonnet esthesiometer

At the 6-weeks visit, participant will be asked to answer a compliance questionnaire.

Treatment The enrolled participants will commence topical application of autologous PRP drops 4 times per day for 6 weeks.

Administration of any other topical medications treating the patient ocular surface will not be allowed during the study period.

ELIGIBILITY:
Inclusion Criteria: Potential participants diagnosed with moderate to sever ocular surface disease. Participant will be included when the fluorescein corne-conjunctival staining score is 5 or more as determined by NEI/Industry Grading System and OSDI questionnaire score of 20 or more, after treatment with non-preserved artificial tears 4/day for at least 1 month.

-

Exclusion Criteria: Under the age of 18 years or incapacitated patients.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Ocular Surface Disease Index (OSDI) score questionnaire | At 6 and 12 weeks visit
  The OSDI assesses quality of life measures of ocular surface disease symptoms which aligns the questionnaire with Federal Food and Drug Administration's emphasis on utilizing patient-reported outcomes in order to support medicinal product submissions and clinical drug trial efficacy

SECONDARY OUTCOMES:
Mean change from baseline of Corneo-conjunctival staining score | At 6 and 12 weeks visit
  Corneo-conjunctival staining scores graded by NEI/Industry Grading System after 1% fluorescein dye staining

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No